CLINICAL TRIAL: NCT04917055
Title: Impact of Adding iPACK Block With Dexamethasone to Existing APS Multimodal Analgesia Protocol for Patients Undergoing Total Knee Arthroplasty
Brief Title: iPACK Block With Dexamethasone For Total Knee Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: staffing
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Engy T. Said, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 210102
Record Dates: First submitted 2021-05-28; First posted 2021-06-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis; Acute Pain; Anesthesia, Local; Regional Anesthesia
Keywords: acute postoperative pain; knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Acute Pain; Pain, Postoperative | interventions — Ropivacaine; Epinephrine; Dexamethasone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Care provider and investigator will know if patient received SHAM or bupivacaine iPACK, but everyone else will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Active Comparator): Adductor Canal Single Shot with long acting local anesthetic (ropivacaine) plus distal iPACK (between femoral condyles) single shot with long acting local anesthetic (ropivacaine) plus dexamethasone
  Interventions: Drug: ropivacaine 0.25% with epinephrine and 6mg dexamethasone
- Placebo (Placebo Comparator): Adductor Canal Single Shot with long acting local anesthetic (ropivacaine) plus iPACK single shot with normal saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: ropivacaine 0.25% with epinephrine and 6mg dexamethasone — Regional Nerve block behind the knee for posterior knee pain following total knee arthroplasty using ultrasound guidance, to be done distally between femoral chondyles
  Arms: Active Treatment
Drug: Saline — Injection of Saline behind knee using ultrasound guidance
  Arms: Placebo

SUMMARY:
Comparing the pain control outcomes for patients undergoing total knee arthroplasty (TKA) with either: 1) adductor canal single shot injection plus placebo iPACK injection or 2) adductor canal single shot injection plus bupivacaine and dexamethasone iPACK injection.

There are two surgical approaches for TKA 1) open 2) ROSA robotic assisted. Both follow the same pain management pathway. We plan to enroll patient undergoing either surgical procedure.

DETAILED DESCRIPTION:
This will be a single-center (UCSD), randomized blinded investigation.

Enrollment. Consenting adults undergoing TKA will be offered enrollment. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current UCSD IRB-approved ICF.

Preoperative Procedures. Following written, informed consent, we will record baseline anthropomorphic information (age, sex, height, and weight) that is already provided by all patients having surgery. After consenting and prior to surgery, patients will be randomized (utilizing sealed envelopes with 1:1 ratio) to either single-shot adductor canal block with sham iPACK block or single-shot adductor canal block with local anesthetic + dexamethasone iPACK block. A regional anesthesia fellow, not participating in the study, will open the sealed envelope and prepare the iPACK solution to be used accordingly.

Current Standard Care: Currently, all patients undergoing TKA receive preoperative adductor canal block as well as multimodal pain regimen managed by APS. They all receive intraoperative intraarticular injections by the surgical team. Spinal vs general anesthesia is decided at the discretion of the intraoperative anesthesiologist along with patient preferences and relevant contraindications. The only difference for subjects participating in the study (vs those not participating) will be that they will be randomized to receive an additional nerve block for posterior knee pain.

Adductor canal single shot block + Sham group: In the preoperative holding area, all subjects in this cohort will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned supine. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion will be cleaned with chlorhexidine gluconate and isopropyl alcohol (ChloraPrep One-Step, Medi-Flex Hospital Products, Inc., Overland Park, KS, USA). A single shot adductor canal block will be performed under ultrasound guidance with 20 mls of 0.25% ropivacaine with 1:400,000 epinephrine. A sensory level to ice will be confirmed and decided to be adequate if positive based on the discretion of the attending anesthesiologist. A Sham iPACK block will then be performed under ultrasound guidance, where 20 mls of 0.9% normal saline with 1:400,000 epi (as a vascular marker) is injected between the popliteal artery and the posterior aspect of the femoral condyle. As is standard for all TKA at our institution, all patients will additionally receive an intraoperative intraarticular injection by the surgical team of 50 mls 0.25% bupivacaine + 30 mg Ketorolac + 0.25mg epinephrine, which will occur at least 60 minutes after preoperative perineural injections.

Adductor canal single shot block + iPACK group: In the preoperative holding area, all subjects in this cohort will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned supine. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion will be cleaned with chlorhexidine gluconate and isopropyl alcohol (ChloraPrep One-Step, Medi-Flex Hospital Products, Inc., Overland Park, KS, USA). A single shot adductor canal block will be performed under ultrasound guidance with 20 mls of 0.25% ropivacaine with 1:400,000 epinephrine. A sensory level to ice will be confirmed and decided to be adequate if positive based on the discretion of the attending anesthesiologist. An iPACK block will then be performed under ultrasound guidance, where 20 mls of 0.25% ropivacaine with 1:400,000 epinephrine and 6mg dexamethasone is injected between the popliteal artery and the posterior aspect of the femoral condyle. As is standard for all TKA at our institution, all patients will additionally receive an intraoperative intraarticular injection by the surgical team of 50 mls 0.25% bupivacaine + 30 mg Ketorolac + 0.25mg epinephrine, which will occur at least 60 minutes after preoperative perineural injections.

Additional Postoperative Pain Interventions: Intraoperatively, spinal anesthesia versus general anesthesia will be decided at the discretion of the operating room anesthesiologist. Postoperatively, both groups will be started on the same multimodal oral regimen and followed by our anesthesiology led acute pain team.

ELIGIBILITY:
Inclusion Criteria:

* Having total knee arthroplasty at UC San Diego
* Plan to receive single shot adductor canal injection preoperatively
* Plan to receive spinal anesthetic with or without sedation for TKA surgery

Exclusion Criteria:

* Pregnancy
* Inability to communicate with anesthesia provider and/or investigators
* Severe renal, hepatic, cardiac disease
* Chronic high-dose opioid use (defined as daily use for more than 4 weeks prior to surgery of at least the equivalent of 20 mg oxycodone)
* BMI > 45 kg/m2
* Allergy to study medications (lidocaine, bupivacaine)
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Average Opioid Use POD 0-1 | Postoperative day (POD) 0-1, as defined by 24 hours after iPACK block placement
  Average Opioid Use
Average Pain Score at Rest | Postoperative day (POD) 0-1, as defined by 24 hours after iPACK block placement
  Average Pain Score at Rest
Average Pain Score with Motion | Postoperative day (POD) 0-1, as defined by 24 hours after iPACK block placement
  Average Pain Score with Motion

SECONDARY OUTCOMES:
Gait Distance | POD0-1 (first PT session)
  Distance patient can walk on with physical therapy (PT)
Knee Range of motion | POD0-1 (first PT session)
  Range of motion with Physical Therapy (PT)
Length of stay | Total number of days requiring hospitalization for surgical procedure. Up to 1 month
  From admission to hospital for surgery to discharge
Average Opioid Use postoperative day (POD) 1-2 | Postoperative day (POD) 1-2.
  Average Opioid Use in morphine equivalents
Average Pain Score, postoperative day (POD) 1-2. | Postoperative day (POD) 1-2.
  Average Pain Score

CONTACTS AND LOCATIONS:
Overall Officials: Engy Said, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No